CLINICAL TRIAL: NCT01415726
Title: Stem Cell Educator Therapy in Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Chinese government (Unknown); Jinan Tianhe Stem Cell Biotechnologies Co Ltd (Unknown)
Responsible Party: Yong Zhao, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-010
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2011-07

CONDITIONS: Type 2 Diabetes
Keywords: Cord blood stem cells; inflammation; type 2 diabetes; stem cell educator; autoimmunity; immune modulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Autoimmune Diseases

ARMS (2):
- Cord blood stem cell (Experimental): Human cord blood-derived multipotent stem cells (CB-SC) display unique phenotypes, such as the expression of embryonic stem (ES) cell markers, multipotential of differentiations, very low immunogenecity, and immune modulations. Stem Cell Educator will be used for isolation and purification of cord blood stem cells for the treatment.
  Interventions: Device: Stem Cell Educator
- Stem Cell Educator (Experimental): used for the isolation and purification of cord blood stem cells.
  Interventions: Device: Stem Cell Educator

INTERVENTIONS:
Device: Stem Cell Educator — For the treatment, commonly the left (or right) median cubital vein, a patient's blood is passed through a Blood Cell Separator that isolates the lymphocytes from the blood according to the recommended protocol by manufacture; consequently, the collected lymphocytes were transferred into the Stem Cell Educator and treated by CB-SC; after that, the educated cells return the blood back to the patient via a dorsal vein of hand. During the MCS+ collection, the whole blood flow rate was maintained at 35 mL/min. The whole procedure was scheduled for 6 ~ 7 hrs.

SUMMARY:
Type 2 diabetes is the most common form of diabetes. The prevalence of diabetes has been markedly increased in recent years. More and more children and young adults develop this devastating disease. Despite of multiple factors (e.g., food, environmental, and genetic factors) contributing to the developing of diabetes, increasing evidence demonstrated that chronic inflammation and/or atuoimmunity are common issues and play key roles in the pathogenesis of type 2 diabetes, leading to the insulin resistance and the shortage of insulin-producing islet beta cells. Thus, anti-inflammation is becoming a novel approach for the treatment of type 2 diabetes. Evidence that multipotent stem cells derived from human cord blood (CB-SCs) can control inflammation and autoimmune responses by altering regulatory T cells (Tregs) and human islet beta cell-specific T cell clone in type 1 diabetes offers promise for a new approach to treat type 2 diabetes. Here, the investigators develop a novel Stem Cell Educator therapy by using CB-SC and explore the therapeutic effectiveness of Stem Cell Educator therapy in T2D patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients were screened for enrollment in the study if both clinical signs and laboratory tests meet the diagnosis standards of American Diabetes Association 2010. Other key inclusion criteria were presence of at least one autoantibody to the pancreatic islet β cells for the autoimmune-related type 2 diabetes.

Exclusion Criteria:

* Exclusion criteria were any clinically significant diseases in liver, kidney, and heart. Additional exclusion criteria were no pregnancy, no immunosuppressive medication, no viral diseases or diseases associated with immunodeficiency.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Inflammation control | 30 days post treatment
  Before treatment, test inflammation-related markers as baseline; After treatment for 30 days, repeat testing inflammation-related markers.

SECONDARY OUTCOMES:
Metabolic control | 3 months
  Before treatment, test for HbA1C levels as baseline; After treatment, test HbA1C levels on the 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhao, MD, PhD, Principal Investigator — Universtiy of Illinois at Chicago
Locations (1):
- General Hospital of Jinan Military Command, Jinan, Shandong, China

REFERENCES:
- [Background] Zhao Y, Mazzone T. Human cord blood stem cells and the journey to a cure for type 1 diabetes. Autoimmun Rev. 2010 Dec;10(2):103-7. doi: 10.1016/j.autrev.2010.08.011. Epub 2010 Aug 20. PMID 20728583
- [Background] Zhao Y, Lin B, Dingeldein M, Guo C, Hwang D, Holterman MJ. New type of human blood stem cell: a double-edged sword for the treatment of type 1 diabetes. Transl Res. 2010 May;155(5):211-6. doi: 10.1016/j.trsl.2010.01.003. Epub 2010 Feb 12. PMID 20403575
- [Background] Zhao Y, Lin B, Darflinger R, Zhang Y, Holterman MJ, Skidgel RA. Human cord blood stem cell-modulated regulatory T lymphocytes reverse the autoimmune-caused type 1 diabetes in nonobese diabetic (NOD) mice. PLoS One. 2009;4(1):e4226. doi: 10.1371/journal.pone.0004226. Epub 2009 Jan 19. PMID 19156219
- [Derived] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Zhou H, Yin Z, Chen Y, Zhang Y, Wang S, Shen J, Thaker H, Jain S, Li Y, Diao Y, Chen Y, Sun X, Fisk MB, Li H. Targeting insulin resistance in type 2 diabetes via immune modulation of cord blood-derived multipotent stem cells (CB-SCs) in stem cell educator therapy: phase I/II clinical trial. BMC Med. 2013 Jul 9;11:160. doi: 10.1186/1741-7015-11-160. PMID 23837842